CLINICAL TRIAL: NCT03235882
Title: Fast Assessment of Surfactant Deficiency to Speed up Treatment: Assessment of Lung Maturity and Prediction of RDS by Determination of L/S-ratio in Fresh Gastric Aspirates by FTIR Spectroscopy
Brief Title: Fast Assessment of Surfactant Deficiency to Speed up Treatment
Acronym: FAST
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Aalborg University Hospital (Other); Aarhus University Hospital (Other); Kolding Sygehus (Other); Odense University Hospital (Other); Herlev Hospital (Other); Hvidovre University Hospital (Other); Holbaek Sygehus (Other)
Responsible Party: Principal Investigator, Christian Heiring, Consultant, Rigshospitalet, Denmark
Other Study IDs: H-17013993
Record Dates: First submitted 2017-07-27; First posted 2017-08-01 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: RDS of Prematurity; Prematurity
Keywords: Lung surfactant; Mid-infrared spectroscopy; Prematurity; Respiratory distress syndrome; gastric aspirate
MeSH Terms: conditions — Respiratory Distress Syndrome In Premature Infants; Premature Birth; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- observational group: Infants born 24-32 weeks.
  Inclusion criteria:
  * Have gastric aspirate and oral secretions obtained within 45 minutes from birth via:
    * a naso- or orogastric tube inserted in the delivery room if clinically indicated as part of resuscitation or
    * a nasogastric tube inserted as part of routine management of preterm infants.
  * Written informed consent has been obtained
  Interventions: Diagnostic Test: LS-ratio

INTERVENTIONS:
Diagnostic Test: LS-ratio — Accurately predict RDS using Lecithin/Sphingomyelin ratio (L/S ratio determined by a rapid FTIR test on fresh gastric aspirates) using retrospective analysis

SUMMARY:
The aim is to validate a FTIR spectroscopy test for measuring lung maturity/Respiratory Distress Syndrome (RDS) in terms of safety, usability, and efficacy.

The purpose is to accurately predict RDS using Lecithin/Sphingomyelin ratio (L/S ratio determined by a rapid FTIR test on fresh gastric aspirates) using retrospective analysis.

Research question:

"In very preterm newborn infants with (risk of) respiratory distress who have not received prophylactic surfactant: does analysis of L/S-ratio in fresh gastric aspirates using a rapid FTIR test predict RDS requiring exogenous surfactant with sufficient specificity and sensitivity to be clinical useful?

DETAILED DESCRIPTION:
Respiratory distress syndrome (RDS) remains a major cause of mortality and morbidity in premature infants despite the increased use of antenatal steroids and early nasal continuous positive airway pressure (nCPAP) in addition to exogenous surfactant replacement therapy(1,2). In recent years, there have been several improvements in treatment, reducing the incidence and severity of RDS and bronchopulmonary dysplasia (BPD) including early treatment with nCPAP, early targeted surfactant replacement therapy, increased used of lung protective ventilation together with an overall reduced use of mechanical ventilation(1,3,4).

However, the majority of premature infants with a gestational age of less than 30 weeks have immature lungs and approximately half still require treatment with exogenous surfactant(2). Timing of surfactant treatment seems crucial. Prophylactic surfactant treatment followed by mechanical ventilation has been widely used, but has now been shown to increase the combined mortality and incidence of BPD, as opposed to early targeted rescue treatment, especially when combined with nCPAP and avoidance of mechanical ventilation using the "Intubation, surfactant, extubation (INSURE) or "Less Invasive Surfactant Administration " (LISA) approach(5-8). In addition, evidence shows that very early targeted surfactant treatment is associated with a better outcome compared to later treatment(9).

Consequently, it is necessary to treat with surfactant selectively and very soon after birth, preferably even before classical symptoms of RDS are present, in order to further improve outcome from RDS. To be able to do so, we need a bedside test that can quickly identify which infants have surfactant deﬁciency to target treatment effectively(1).

Biomarkers expressing lung maturity have been identiﬁed in amniotic ﬂuid, gastric aspirate, and oropharyngeal secretions(10-12). These ﬂuids are partially produced in the foetal lungs as well as in the kidneys and the amniotic sac and therefore contain lung surfactant(13). The classic method to determine surfactant in amniotic ﬂuid has been measuring lecithin/sphingomyelin ratio (L/S) with thin-layer chromatography(10,14). Sphingomyelin secretion remains fairly constant during pregnancy, whereas lecithin secretion increases in parallel with lung maturation. Consequently, L/S-ratio reﬂects lung maturity independently of dilution sampling effects(10)

Gastric aspirate (GAS) and oropharyngeal (OPS) secretion are easier to obtain and measure than amniotic ﬂuid, and can be obtained within minutes from birth using routine neonatal care measures(15,16). Previously, we have measured the surfactant content in gastric aspirate with microbubble stability tests and with lamellar body counts(17,18). In a recent randomized clinical trial in very preterm infants we compared early surfactant treatment guided by lamellar body counts in gastric aspirate with traditional surfactant treatment, and found a significant reduction in the need of oxygen at six hours of age and by day 28, in addition to reduced duration of oxygen-dependency and a trend towards a lower incidence of bronchopulmonary dysplasia(19).

However, both the microbubble stability test and lamellar body counts are work and laboratory intensive and require a minimum of two to three hours for analysis.

The investigators have developed a fast method based on Fourier Transform Infrared (FTIR) Spectroscopy for determining the L/S ratio in gastric aspirate and secretion from the oropharynx. In a recent study, the algorithms for FTIR L/S analyses were developed and improved 20). Concentrations were measured of the most surface-active lung phospholipid dipalmitoylphosphatidylcholine and sphingomyelin in frozen gastric aspirates from 89 premature infants expressed as lecithin/sphingomyelin ratio (L/S) by mass spectrometry as the reference method. The same aspirates were analyzed with FTIR spectroscopy. An L/S algorithm was developed based on the 89 aspirates. Subsequently gastric aspirates were sampled in 136 infants of 24-31 weeks of gestation. L/S was measured in these frozen gastric aspirates using FTIR spectroscopy and the results were compared with RDS development. Of 136 infants 61 (45%) developed RDS. The cut-off value of L/S was 2.2, sensitivity was 92% and specificity was 73%. The FTIR spectroscopy analysis required 10 μL of aspirate and took 10 minutes.

In an effort to increase accuracy and reproducibility, the investigators have continued to improve the FTIR spectroscopy method and algorithms by making comparative measurements with mass spectrometry using fresh non-frozen aspirates from newborn infants. These improvements may also have affected the optimal cut-off value in our test.

The investigators are in the process of planning a large multicenter randomized clinical trial of FTIR spectroscopy guided surfactant treatment using a point of care (POC) device based on the FTIR algorithms and techinique using fresh aspirates that can be analyzed immidiately in birth suite or the NICU. Before embarking on an interventional study however, it is needed to re-validate the updated and improved FTIR spectroscopy test by again comparing clinical appearance of RDS with L/S-ratio measured by FTIR spectroscopy on fresh non-frozen gastric aspirates froma new population of preterm infants.

Hypothesis: Fast determination of Lecithin/Sphingomyelin-ratio (L/S-ratio) in gastric aspirates by FTIR Spectroscopy, can accurately and consistently predict RDS based on clinical criteria.

Trial design The trial is designed as prospective non-intervention observational cohort study, with the aim to assess the efficacy in predicting RDS by a LS-test on fresh gastric aspirates and oral secretions based on FTIR spectroscopy, by comparing clinical progress with the LS-ratio. Included infants will be treated according to routine guidelines and at the discretion of the attending neonatologist. No interventions are planned to be based on the result of the L/S test.

AMMENTMENT:

We have ammended the project with an attempt to use the same method and AI combined with clinical data to predict development of BPD, defined as continued requirements for supplemental oxygen to DOL28. Spectroscopic measurements were done again using stored gastric aspirate from the first part of the study.

This amendment has been approved by HREC and measurements were only done after parents gave informed consent for participation of this additional part of the study.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria:

* Have GAS obtained within 45 minutes from birth via:

  * a naso- or orogastric tube inserted in the delivery room if clinically indicated as part of resuscitation or
  * a nasogastric tube inserted as part of routine management of preterm infants.
* Written informed consent has been obtained

Exclusion Criteria:

* Intubated and treated with surfactant before obtaining GAS
* Diagnosis of lethal malformations
* Antenatal diagnosis of lung hypoplasia
* Therapeutic infusion given in the amniotic cavity
* GAS unavailable or significantly contaminated by meconium/pus
* Sepsis

Max Age: 45 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm newborn babies that have gastric/oral secretions sampled before 45 minutes of age
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
development of RDS | 5 days from delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neonatology, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Publication of the completed study — https://www.ncbi.nlm.nih.gov/pubmed/31038796